CLINICAL TRIAL: NCT06094751
Title: Online ACT Guide for Sub-clinical and Clinical Insomnia Among College Students
Brief Title: An ACT Website for College Students With Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Twohig, Ph.D., Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13376
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Insomnia
Keywords: Insomnia; college student; university student; online
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Guide for Insomnia (Experimental): Participants will complete 2 modules of an online Acceptance and Commitment Therapy (ACT) Guide designed to focus on insomnia among college students. Module 1 will be available to participants at the start of week 1 and throughout the course of the study. Module 2 will become available at the start of week 3 and participants will have access throughout the study
  Interventions: Behavioral: ACT Guide for Insomnia
- Waitlist (No Intervention): Participants randomized into the waitlist condition will not have access to the ACT Guide for Insomnia until the conclusion of their time in the study (8 weeks after randomization).

INTERVENTIONS:
Behavioral: ACT Guide for Insomnia — ACT Guide for Insomnia includes 2 modules. Module 1 will include sleep/insomnia education, ACT skills (acceptance, defusion), and behavioral change. Module 2 will include sleep restriction, sleep hygiene, ACT skills (values, committed action), and behavioral change.
  Arms: ACT Guide for Insomnia

SUMMARY:
College students experience higher rates of insomnia compared the general population, and accessibility and availability for the appropriate intervention is difficult due limited resources available to them in a college environment. Theorefore, it is vital to offer an intervention that can be just as effective yet more accessible than other available treatments targeting insomnia. That is why this study will investigate the efficacy and feasibility of an online ACT intervention for insomnia among college students. Specifically, Is an online ACT for college students effective in treating insomnia? And, is an online ACT for college students feasible and acceptable in treating insomnia? Participants will be randomized into one of two conditions: waitlist or online ACT guide. Participants will receive questionnaires at baseline, post-treatment (4 weeks), and 1-month follow up.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. enrolled in a 2- or 4-year college (includes graduate students)
3. fluent in English
4. have access to the internet
5. meets diagnosis for at least acute insomnia according to the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5
6. searching/wanting in treatment
7. currently residing in the US

Exclusion Criteria:

1. diagnosed with another sleep disorder that is not insomnia
2. currently attending therapy for an emotional disorder (anxiety or depression) or insomnia
3. prescribed medications to treat insomnia or another sleep-inducing medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 8 weeks
  The ISI is composed of 7-items that asses for severity of sleep onset, sleep maintenance, early morning waking issues, sleep satisfaction, sleep interference (e.g., daytime fatigue), noticeability of sleep impairment, and sleep worry. Each item is measured on a five-point likert scale ranging from 0 indicating no severity to 4 indicating very severe. The ISI has been shown to be a valid, clinical questionnaire designed to gauge insomnia severity (Bastien, Vallières, & Morin, 2001), is sensitive to treatment response (Morin, Belleville, Bélanger, & Ivers, 2011), and has been agreed upon as essential for insomnia treatment efficacy studies (Buysse, Ancoli-Israel, Edinger, Lichstein, & Morin, 2006). Additionally, the ISI has been used a previous randomized control trails (RCT) among college student to determine treatment efficacy (Taylor et al., 2014).

CONTACTS AND LOCATIONS:
Locations (1):
- Utah State University, Logan, Utah, United States